CLINICAL TRIAL: NCT03055156
Title: Effect of High Rebound Mattress Toppers on Sleep and Sleep-Related Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Airweave Pte Ltd. (Industry)
Responsible Party: Principal Investigator, Seiji Nishino, Professor, Psychiatry and Behavioral Sciences, Stanford University School of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB-34797
Record Dates: First submitted 2015-08-26; First posted 2017-02-16 (Actual); Results first posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-10

CONDITIONS: Sleep Disorders
Keywords: Sleep Apnea; Insomnia; sleep disorders; sleep environment; core body temperature
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Apnea Syndromes; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Low rebound mattress toppers (Experimental): sleep with mattress topper during overnight diagnostic sleep study
  Interventions: Device: Low rebound mattress toppers
- High rebound mattress toppers (Experimental): sleep with mattress topper during overnight diagnostic sleep study
  Interventions: Device: High rebound mattress toppers

INTERVENTIONS:
Device: Low rebound mattress toppers — Patients will sleep on this mattress topper during their diagnostic sleep study.
  Other Names: TEMPUR-Topper Supreme
  Arms: Low rebound mattress toppers
Device: High rebound mattress toppers — Patients will sleep on this mattress topper during their diagnostic sleep study.
  Other Names: airweave® mattress topper
  Arms: High rebound mattress toppers

SUMMARY:
The purpose of the study is to evaluate effects of high rebound mattress toppers (i.e., airweave®) on sleep and sleep-related symptoms.

The study will compare effects of use of high rebound mattress toppers versus use of low rebound mattress toppers on sleep and sleep related symptoms and core body temperature during diagnostic sleep studies.

ELIGIBILITY:
Inclusion Criteria:

* Adults Age 18-65 who are scheduled for a diagnostic sleep study at the Stanford Sleep Clinic for sleep disorders (including but not limited to, insomnia, Sleep Apnea or other sleep disorder symptoms).

Exclusion Criteria:

* Individuals with a history of having difficulty swallowing food or large capsules. We will not be able to enroll individuals with any known or suspected obstructive disease of the gastrointestinal tract including, but not limited to esophageal stricture, diverticulosis and inflammatory bowel disease (IBD), peptic ulcer disease, Crohn's disease, ulcerative colitis, previous gastrointestinal surgery.
* Individuals who are pregnant.
* Individuals who are unable to provide informed consent (i.e. decisionally impaired).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2015-10; Primary Completion 2019-10-19 (Actual); Study Completion 2019-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seiji Nishino, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford Sleep Research Center, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from individuals who were scheduled for an overnight PSG study as part of their regular care at the Stanford Sleep clinic.
Pre-assignment Details: 4 participants were enrolled but not randomized to a study arm.
Groups:
- Low Rebound Mattress Toppers: Participants in arm 1 slept on low rebound mattress toppers (Topper Deluxe 3.5, TEMPUR-SEALY Japan Ltd., Kobe, Japan) placed on top of standard mattresses equipped at the Stanford Sleep Clinic.
- High Rebound Mattress Toppers: Participants in arm 2 slept on high rebound mattress toppers (airweave® toppers, airweave inc., Tokyo, Japan) placed on top of standard mattresses equipped at the Stanford Sleep Clinic.
Period: Overall Study
Arm/Group | Low Rebound Mattress Toppers | High Rebound Mattress Toppers
Started | 281 | 273
Completed | 281 | 273
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- Low Rebound Mattress Toppers: Participants in arm 1 slept on low rebound mattress toppers placed on top of standard mattresses equipped at the Stanford Sleep Clinic.
- High Rebound Mattress Toppers: Participants in arm 2 slept on high rebound mattress toppers placed on top of standard mattresses equipped at the Stanford Sleep Clinic.
- Total: Total of all reporting groups
Arm/Group | Low Rebound Mattress Toppers | High Rebound Mattress Toppers | Total
Number analyzed (Participants) | 281 | 273 | 554
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age was collected through online form, and not all participants entered age information.
  years
    number analyzed (Participants) | 200 | 175 | 375
    (all) | 39.42 (15.84) | 41.27 (15.93) | 40.28 (15.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 135 | 264
  Male | 152 | 138 | 290
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 44 | 42 | 86
  Black/African American | 8 | 14 | 22
  Hispanic/Latino | 18 | 26 | 44
  Native Hawaiian/Pacific Islander | 1 | 2 | 3
  Native American | 2 | 0 | 2
  White/Caucasian | 186 | 173 | 359
  Multiple | 7 | 4 | 11
  Unknown | 1 | 0 | 1
  Other | 7 | 12 | 19
  Participant indicated Multiple and Other | 7 | 2 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 281 | 273 | 554
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.22 (5.61) | 26.34 (5.41) | 26.30 (5.51)
Room temperature [Mean (Standard Deviation); unit: degrees Celsius] — Population: Room temperature was not recorded for all participants.
  degrees Celsius
    number analyzed (Participants) | 215 | 215 | 430
    (all) | 20.84 (1.41) | 20.88 (1.42) | 20.84 (1.41)

OUTCOME MEASURES:

1. Primary Outcome: Total Sleep Time
Time Frame: Overnight study visit (up to approximately 10hrs)
Population: Participants with non missing data, who completed the study during the night, and did not initiate CPAP or biPAP during the study were included in the analysis.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Low Rebound Mattress Toppers | High Rebound Mattress Toppers
Number analyzed (Participants) | 216 | 200
hours | 6.62 (1.25) | 6.55 (1.59)
Statistical Analysis 1: Comparison: Low Rebound Mattress Toppers vs High Rebound Mattress Toppers; Test type: Other; p = 0.60, t-test, 2 sided

2. Primary Outcome: Sleep Efficiency Assessed by Polysomnography (PSG)
Description: Sleep efficiency is total sleep time divided by time in bed. All data were collected through the PSG data that were retrieved from the patients' medical records after completion of the recordings and analysis by the sleep technologists.
Time Frame: Overnight study visit (up to approximately 10hrs)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage time in bed asleep
Arm/Group | Low Rebound Mattress Toppers | High Rebound Mattress Toppers
Number analyzed (Participants) | 216 | 200
percentage time in bed asleep | 82.87 (11.34) | 79.73 (14.94)
Statistical Analysis 1: Comparison: Low Rebound Mattress Toppers vs High Rebound Mattress Toppers; Test type: Other; p = 0.02, t-test, 2 sided

3. Primary Outcome: Sleep Latency Assessed by PSG
Description: The amount of time from lights off to falling asleep.
Time Frame: Overnight study visit (up to approximately 10hrs)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Low Rebound Mattress Toppers | High Rebound Mattress Toppers
Number analyzed (Participants) | 214 | 199
minutes | 18.67 (21.00) | 24.05 (25.31)
Statistical Analysis 1: Comparison: Low Rebound Mattress Toppers vs High Rebound Mattress Toppers; Test type: Other; p = 0.02, t-test, 2 sided

4. Primary Outcome: Wake After Sleep Onset (WASO) Assessed by PSG
Description: Total amount of minutes awake after the first sleep epoch.
Time Frame: Overnight study visit (up to approximately 10hrs)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Low Rebound Mattress Toppers | High Rebound Mattress Toppers
Number analyzed (Participants) | 215 | 199
minutes | 60.09 (43.57) | 74.36 (67.55)
Statistical Analysis 1: Comparison: Low Rebound Mattress Toppers vs High Rebound Mattress Toppers; Test type: Other; p = 0.01, t-test, 2 sided

5. Primary Outcome: Percentage of Time in Bed During Each Sleep Stage
Time Frame: Overnight study visit (up to approximately 10hrs)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of time in bed
Arm/Group | Low Rebound Mattress Toppers | High Rebound Mattress Toppers
Number analyzed (Participants) | 214 | 198
percentage of time in bed
  Wake | 17.11 (11.38) | 20.16 (14.92)
  REM | 16.26 (6.96) | 14.92 (7.52)
  Non REM stage 1 | 6.36 (4.83) | 6.46 (4.58)
  Non REM stage 2 | 47.67 (12.22) | 47.36 (12.69)
  Non REM stage 3 | 11.86 (10.58) | 11.81 (16.09)
Statistical Analysis 1: Comparison: Low Rebound Mattress Toppers vs High Rebound Mattress Toppers; Analysis of Wake values; Test type: Other; p = 0.02, t-test, 2 sided
Statistical Analysis 2: Comparison: Low Rebound Mattress Toppers vs High Rebound Mattress Toppers; Analysis of REM values; Test type: Other; p = 0.06, t-test, 2 sided
Statistical Analysis 3: Comparison: Low Rebound Mattress Toppers vs High Rebound Mattress Toppers; Analysis of Non REM stage 1 values; Test type: Other; p = 0.83, t-test, 2 sided
Statistical Analysis 4: Comparison: Low Rebound Mattress Toppers vs High Rebound Mattress Toppers; Analysis of Non REM stage 2 values; Test type: Other; p = 0.87, t-test, 2 sided
Statistical Analysis 5: Comparison: Low Rebound Mattress Toppers vs High Rebound Mattress Toppers; Analysis of Non REM stage 3 values; Test type: Other; p = 0.97, t-test, 2 sided

6. Primary Outcome: Position Changes Assessed by PSG
Description: Number of times participant changed position during the sleep recording.
Time Frame: Overnight study visit (up to approximately 10hrs)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of position changes
Arm/Group | Low Rebound Mattress Toppers | High Rebound Mattress Toppers
Number analyzed (Participants) | 213 | 197
number of position changes | 14.64 (12.76) | 15.65 (10.45)
Statistical Analysis 1: Comparison: Low Rebound Mattress Toppers vs High Rebound Mattress Toppers; Test type: Other; p = 0.38, t-test, 2 sided

7. Primary Outcome: Apnea Hypopnea Index Assessed by PSG
Description: The number of apneas or hypopneas recorded during the study per hour of sleep.
Time Frame: Overnight study visit (up to approximately 10hrs)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of events per hour
Arm/Group | Low Rebound Mattress Toppers | High Rebound Mattress Toppers
Number analyzed (Participants) | 213 | 198
number of events per hour | 34.15 (57.00) | 33.86 (45.48)
Statistical Analysis 1: Comparison: Low Rebound Mattress Toppers vs High Rebound Mattress Toppers; Test type: Other; p = 0.96, t-test, 2 sided

8. Primary Outcome: Heart Rate
Time Frame: Overnight study visit (up to approximately 10hrs)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Low Rebound Mattress Toppers | High Rebound Mattress Toppers
Number analyzed (Participants) | 216 | 200
Beats per minute | 61.24 (14.19) | 64.82 (10.48)

9. Primary Outcome: Periodic Leg Movements (PLM) During Sleep
Description: Number of times participant had periodic leg movements during the sleep recording
Time Frame: Overnight study visit (up to approximately 10hrs)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of PLM events
Arm/Group | Low Rebound Mattress Toppers | High Rebound Mattress Toppers
Number analyzed (Participants) | 203 | 181
number of PLM events | 99.56 (143.43) | 91.51 (11.36)
Statistical Analysis 1: Comparison: Low Rebound Mattress Toppers vs High Rebound Mattress Toppers; Test type: Other; p = 0.55, t-test, 2 sided

10. Primary Outcome: Mean EEG Delta Spectral Power Per Second Over 90 Mins From Lights Off Between 0-360 Minutes After Lights Off
Description: EEG data collected from the electrode in position C2
Time Frame: Overnight study visit (up to approximately 10hrs)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µV^2
Arm/Group | Low Rebound Mattress Toppers | High Rebound Mattress Toppers
Number analyzed (Participants) | 210 | 196
µV^2
  0-90min | 31.34 (30.71) | 31.93 (36.61)
  90-180min | 28.61 (31.56) | 32.00 (32.61)
  180-270min | 24.19 (31.55) | 27.02 (67.62)
  270-360min: number analyzed (Participants) | 209 | 195
  270-360min | 21.66 (38.68) | 20.07 (23.35)
Statistical Analysis 1: Comparison: Low Rebound Mattress Toppers vs High Rebound Mattress Toppers; analysis of 0-90 minutes; Test type: Other; p = 0.86, t-test, 2 sided
Statistical Analysis 2: Comparison: Low Rebound Mattress Toppers vs High Rebound Mattress Toppers; analysis of 90-180 minutes; Test type: Other; p = 0.29, t-test, 2 sided
Statistical Analysis 3: Comparison: Low Rebound Mattress Toppers vs High Rebound Mattress Toppers; analysis of 180-270 minutes; Test type: Other; p = 0.58, t-test, 2 sided
Statistical Analysis 4: Comparison: Low Rebound Mattress Toppers vs High Rebound Mattress Toppers; analysis of 270-360 min; Test type: Other; p = 0.62, t-test, 2 sided

11. Secondary Outcome: Core Body Temperature
Description: Difference in core body temperature changes of the high and low rebound mattress toppers at sleep onset and during sleep. The core body temperature will be monitored every minute throughout the night.
Time Frame: Overnight study visit (up to approximately 10hrs)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | Low Rebound Mattress Toppers | High Rebound Mattress Toppers
Number analyzed (Participants) | 145 | 142
degrees Celsius
  30min since lights off | 36.42 (1.15) | 36.29 (1.23)
  60min since lights off | 36.49 (0.34) | 36.52 (0.34)
  90min since lights off | 36.46 (0.34) | 36.49 (0.35)
  120min since lights off | 36.47 (0.33) | 36.51 (0.34)
  150min since lights off | 36.51 (0.33) | 36.53 (0.32)
  180min since lights off | 36.54 (0.32) | 36.56 (0.31)
  210min since lights off | 36.56 (0.33) | 36.57 (0.30)
  240min since lights off | 36.59 (0.31) | 36.61 (0.32)
  270min since lights off | 36.58 (0.36) | 36.64 (0.38)
  300min since lights off | 36.59 (0.33) | 36.65 (0.30)
  330min since lights off | 36.61 (0.28) | 36.64 (0.29)
  360min since lights off | 36.62 (0.28) | 36.63 (0.29)
Statistical Analysis 1: Comparison: Low Rebound Mattress Toppers vs High Rebound Mattress Toppers; Implemented two-way mixed ANOVA with time as within-subject variable and topper type as between-subject variable. This is to compare the difference in core body temperature trend over time between the two study arms. Interaction between time and topper type on CBT was calculated; Test type: Other; p = 0.389, ANOVA
Statistical Analysis 2: Comparison: Low Rebound Mattress Toppers vs High Rebound Mattress Toppers; Implemented two-way mixed ANOVA with time as within-subject variable and topper type as between-subject variable. This is to see the effect over time from both study arms on CBT. Main effect of time on CBT; Test type: Other; p = 0.01, ANOVA
Statistical Analysis 3: Comparison: Low Rebound Mattress Toppers vs High Rebound Mattress Toppers; Implemented two-way mixed ANOVA with time as within-subject variable and topper type as between-subject variable. This is to see the effect of the intervention on CBT including all time points. Main effect of topper type on CBT; Test type: Other; p = 0.642, ANOVA

12. Secondary Outcome: Visual Analog Scale of Sleep
Description: visual analog scale of sleep was used for evaluation of subjective sleep quality. Scale ranged from 0 cm (very bad) to 10 cm (very good).
Time Frame: Overnight study visit (up to approximately 10hrs)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Rebound Mattress Toppers | High Rebound Mattress Toppers
Number analyzed (Participants) | 194 | 170
units on a scale | 4.93 (2.33) | 4.80 (2.45)
Statistical Analysis 1: Comparison: Low Rebound Mattress Toppers vs High Rebound Mattress Toppers; Test type: Other; p = 0.61, t-test, 2 sided

13. Secondary Outcome: Visual Analog Scale of Performance
Description: visual analog scale of performance was used for evaluation of subjective performance quality. Scale ranged from 0 cm (very bad) to 10 cm (very good).
Time Frame: Overnight study visit (up to approximately 10hrs)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Rebound Mattress Toppers | High Rebound Mattress Toppers
Number analyzed (Participants) | 192 | 167
units on a scale | 5.54 (2.21) | 5.45 (2.35)
Statistical Analysis 1: Comparison: Low Rebound Mattress Toppers vs High Rebound Mattress Toppers; Test type: Other; p = 0.71, t-test, 2 sided

14. Secondary Outcome: Visual Analog Scale of Mood
Description: visual analog scale of mood was used for evaluation of subjective mood. Scale ranged from 0 cm (very bad) to 10 cm (very good).
Time Frame: Overnight study visit (up to approximately 10hrs)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Low Rebound Mattress Toppers | High Rebound Mattress Toppers
Number analyzed (Participants) | 192 | 169
units on a scale | 6.60 (2.06) | 6.60 (2.03)
Statistical Analysis 1: Comparison: Low Rebound Mattress Toppers vs High Rebound Mattress Toppers; Test type: Other; p = 1.00, t-test, 2 sided

15. Secondary Outcome: Alliance Sleep Questionnaire (ASQ)
Description: self-reported information related to sleep
Time Frame: Overnight study visit (up to approximately 10hrs)
Population: Data were not collected for this outcome measure.
Arm/Group | Low Rebound Mattress Toppers | High Rebound Mattress Toppers
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Study visit overnight (up to 24hrs)
Arm/Group | Low Rebound Mattress Toppers | High Rebound Mattress Toppers
All-Cause Mortality (participants affected / at risk) | 0/281 | 0/273
Serious Adverse Events (participants affected / at risk) | 0/281 | 0/273
Other Adverse Events (participants affected / at risk) | 0/281 | 0/273

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2015-08-04): https://cdn.clinicaltrials.gov/large-docs/56/NCT03055156/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-13): https://cdn.clinicaltrials.gov/large-docs/56/NCT03055156/SAP_001.pdf